CLINICAL TRIAL: NCT05237843
Title: Hydroxychloroquine in Unexplained Recurrent Pregnancy Loss ,Double Blinded Randomized Controlled Trial .
Brief Title: Hydroxychloroquine in Unexplained Recurrent Pregnancy Loss
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HCQ in URPL
Record Dates: First submitted 2021-11-23; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Pregnancy Loss
MeSH Terms: interventions — Hydroxychloroquine; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: Group A (control group) : 35 women in this group will receive only the standard treatment in the form of low- dose aspirin (LDA) 81 mg/day (Jusprin® 81mg which manufactured by Future Pharmaceutical Company), and LMWH (Enoxaparin, Clexane® which manufactured by SANOFI company) with a dose ( .5 mg/kg) subcutaneously injected/24 hr . LDA ought to be begun before origination, while LMWH ought to be begun after confirmation of pregnancy by detecting fetal viability by ultrasound plus Placebo specially manufactured tablets in our Ain shams faculty of pharmacy .
  Group B ( Hydroxychloroquine group ) : This group included 35 women who will administered Hydroxychloroquine 200 mg (Hydroquine® 200mg which fabricated by MinaPharm Company) one tablets / day in addition to the standard therapy
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each 70 sequential patient numbers were composed murky envelope while task code composed different paper that then fixed inside. At hour predisposition visit individual control opened envelope to uncover task, continued like manner (bunch A or B ).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (control group) (Placebo Comparator): 35 women in this group will receive only the standard treatment in the form of :
  * low- dose aspirin (LDA) 81 mg/day orally (Jusprin® 81mg which manufactured by Future Pharmaceutical Company),
  * LMWH (Enoxaparin, Clexane® which manufactured by SANOFI company) with a dose ( .5 mg/kg) subcutaneously injected/24 hr .
  LDA ought to be begun before origination, while LMWH ought to be begun after confirmation of pregnancy by detecting fetal viability by ultrasound till age of viability (20wks)
  -PLUS Placebo specially manufactured tablets in Ain shams faculty of pharmacy will start once known she is pregnan
  Interventions: Drug: Hydroxychloroquine
- Group B ( Hydroxychloroquine group ) (Experimental): This group included 35 women who will administered Hydroxychloroquine 200 mg (Hydroquine® 200mg which fabricated by MinaPharm Company) one tablets / day once known she is pregnant in addition to the standard therapy (LMWH + LDA )
  Interventions: Drug: Hydroxychloroquine
- Study Director (No Intervention): Only those directing the study know the treatment that each participant receives Placebo OR Hydroxychloroquin

INTERVENTIONS:
Drug: Hydroxychloroquine — Besides anti-thrombotic effects, hydroxychloroquine have immunoregulatory properties and can block the production of pro-inflammatory cytokines ( Mekinian A et al ,2015 ) , Few in vitro studies showed a potential benefit of hydroxychloroquine in early trophoblastic migration and implantation. Hydroxychloroquine restored trophoblastic fusion and differentiation and restored the annexin A5 expression.( Guller S et al ,2011 )
  Other Names: placebo - Aspirin (LDA) - Clexan (LMWH)
  Arms: Group A (control group); Group B ( Hydroxychloroquine group )

SUMMARY:
To investigate efficacy and safety of Hydroxychloroquin in improving pregnancy outcome in women with unexplained recurrent pregnancy loss .

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL) remains a significant challenge in obstetrical practice. It is not only emotionally devastating for expectant women but is also medically challenging. Approximately 1-3% of women have recurrent spontaneous abortion, defined as ≥3 pregnancy losses before the age of viability .The European Society of Human Reproduction and Embryology (ESHRE 2021) defined RPL as three or more consecutive losses. The American College of Obstetrics and Gynecology (ACOG 2020) defined RPL as two or more consecutive losses and the American Society for Reproductive Medicine (ASRM 2021) defined RPL as two or more failed pregnancies.

RPL maybe due to uterine anatomic anomalies, endocrine/hormonal abnormalities, genetic/chromosomal abnormalities, and blood coagulation/platelet defects . Many of these causes are treatable . However, in about 40%-50% of pregnancy-loss cases, there is no identifiable cause. As such, the term "unexplained recurrent pregnancy loss" (URPL) is the spontaneous loss of three or more consecutive pregnancies without an identifiable risk factor .

Endometrial environment plays a crucial place in embryo implantation and early placental development. In normal pregnancy, the survival of the semi-allogeneic fetus is dependent on the induction of maternal immune tolerance, with decrease regulatory T cells and Th-2 anti-inflammatory profile in peripheral blood and endometrium .

Several reports show a misbalance of immune cells and cytokines expression such as increased Th1 to Th2 cytokine ratio in women with recurrent miscarriage and implantation failure .The excess activation of the proinflammatory pathways may inhibit the proliferation and invasion of the extravillous trophoblast and induce the activation of the immune cells with a direct damage to the trophoblast . So several studies have highlighted the immune deregulation to explain URM , Consequently, it has been hypothesized that immunomodulatory drugs could be a relevant therapy in URM .Among them, various treatments have been recently used, as HCQ . .

Heparin-based drugs are essential in treating thrombosis and embolisms and preventing thromboembolic phenomena. Heparin works primarily by inhibiting thrombin (factor IIa) and factor Xa. Heparin use is associated with the risk of bleeding, osteoporosis and heparin-induced thrombocytopenia so requiring close monitoring .Apart from its antithrombotic effects, heparin has anti-inflammatory effect which consist to prevent the endothelial cells adhesion to the endothelium; heparin can bind selectins and integrins and interfere with complement activation. But these anti-thrombotic treatments have been used for several years to enhance live birth rates in URM, but failed to reach significant efficacy .

Besides anti-thrombotic effects, hydroxychloroquine have immunoregulatory properties and can block the production of pro-inflammatory cytokines , Few in vitro studies showed a potential benefit of hydroxychloroquine in early trophoblastic migration and implantation. Hydroxychloroquine restored trophoblastic fusion and differentiation and restored the annexin A5 expression .

Hydroxychloroquine is widely used during the pregnancy, in particular in patients with systemic lupus erythematous. The main severe adverse effects in mothers include the allergic reactions, potential heart toxicity, and retinopathy. The retinal toxicity mainly concerns treatment duration of more than 5 years and the risk remain low in patients with regular follow-up . Audio-vestibular and ophthalmological studies of children at 12 months of life born from mothers under hydroxychloroquine during pregnancy showed no apparent abnormality and were similar to non-exposed children.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 35 years inclusive.
* Women with at least three previous consecutive miscarriages in the first trimester of pregnancy of unknown origin with no uterine cavity abnormality that might explain recurrent miscarriage at 3D ultrasonography
* Women who have given their informed consent.
* Patient who did received standard treatment and failed in an ongoing pregnancy

Exclusion Criteria:

* Previous history VTE (venous thromboembolization)
* Persistent positive APL antibodies: lupus anticoagulant and/or APL (anticardiolipin or anticardiolipin IgG or IgM) titers >99th percentile or >40 with at least 12 weeks interval between two positive determinations (persistent antibodies) or a specific clinical setting of APS (thrombotic or obstetrical, apart from RM in the first trimester of pregnancy) .
* Known contraindication to a treatment by HCQ (retinopathy, hypersensitivity to chloroquine or HCQ, G6PD deficiency, acute intermittent porphyria, chronic liver or kidney insufficiency, extensive cutaneous psoriasis not controlled by local treatment, significant chronic digestive or haematologic disease) .
* Indication to a treatment by HCQ (rheumatoid arthritis, Lupus, solar eczema) or previous exposure for >5years to HCQ.
* BMI > 35
* Condition may have an effect on immune reaction e.g. history of HCV or HBV .
* Endocrinopathies such as ( DM ,thyroid disorders , hyperprolactinemia ) .
* History of hormonal contraception or intrauterine device usage in last 3 months preceeding .

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — study will go on pregnant females
Enrollment: 70 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
To investigate HCQ as a new edition in URPL protocol in change rate of pregnancy loss side by side with anticoagulant traditional treatment | one year to be completed
  Describing 200 mg of HCQ daily in unexplained recurrent pregnancy loss start once she makes sure of pregnancy till 20 weeks of pregnancy

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to new guide for recurrent pregnancy lss. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party
Supporting Information: Study Protocol, CSR
Time Frame: Basline
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact: yasmineabdoud@gmail.com

REFERENCES:
- [Result] Alijotas-Reig J, Garrido-Gimenez C. Current concepts and new trends in the diagnosis and management of recurrent miscarriage. Obstet Gynecol Surv. 2013 Jun;68(6):445-66. doi: 10.1097/OGX.0b013e31828aca19. PMID 23942472
- [Result] de Jong PG, Kaandorp S, Di Nisio M, Goddijn M, Middeldorp S. Aspirin and/or heparin for women with unexplained recurrent miscarriage with or without inherited thrombophilia. Cochrane Database Syst Rev. 2014 Jul 4;2014(7):CD004734. doi: 10.1002/14651858.CD004734.pub4. PMID 24995856
- [Result] Sperber K, Hom C, Chao CP, Shapiro D, Ash J. Systematic review of hydroxychloroquine use in pregnant patients with autoimmune diseases. Pediatr Rheumatol Online J. 2009 May 13;7:9. doi: 10.1186/1546-0096-7-9. PMID 19439078
- [Result] Garrido-Gimenez C, Alijotas-Reig J. Recurrent miscarriage: causes, evaluation and management. Postgrad Med J. 2015 Mar;91(1073):151-62. doi: 10.1136/postgradmedj-2014-132672. Epub 2015 Feb 13. PMID 25681385
- [Result] Duckitt K, Qureshi A. Recurrent miscarriage. BMJ Clin Evid. 2011 Feb 1;2011:1409. PMID 21718553
- [Result] Alijotas-Reig J, Llurba E, Gris JM. Potentiating maternal immune tolerance in pregnancy: a new challenging role for regulatory T cells. Placenta. 2014 Apr;35(4):241-8. doi: 10.1016/j.placenta.2014.02.004. Epub 2014 Feb 14. PMID 24581729
- [Result] Liang PY, Diao LH, Huang CY, Lian RC, Chen X, Li GG, Zhao J, Li YY, He XB, Zeng Y. The pro-inflammatory and anti-inflammatory cytokine profile in peripheral blood of women with recurrent implantation failure. Reprod Biomed Online. 2015 Dec;31(6):823-6. doi: 10.1016/j.rbmo.2015.08.009. Epub 2015 Aug 21. PMID 26371706
- [Result] Lim KJ, Odukoya OA, Ajjan RA, Li TC, Weetman AP, Cooke ID. The role of T-helper cytokines in human reproduction. Fertil Steril. 2000 Jan;73(1):136-42. doi: 10.1016/s0015-0282(99)00457-4. PMID 10632428
- [Result] Otun HA, Lash GE, Innes BA, Bulmer JN, Naruse K, Hannon T, Searle RF, Robson SC. Effect of tumour necrosis factor-alpha in combination with interferon-gamma on first trimester extravillous trophoblast invasion. J Reprod Immunol. 2011 Jan;88(1):1-11. doi: 10.1016/j.jri.2010.10.003. Epub 2010 Nov 26. PMID 21112094
- [Result] Haddad EK, Duclos AJ, Antecka E, Lapp WS, Baines MG. Role of interferon-gamma in the priming of decidual macrophages for nitric oxide production and early pregnancy loss. Cell Immunol. 1997 Oct 10;181(1):68-75. doi: 10.1006/cimm.1997.1199. PMID 9344498
- [Result] Onishi A, St Ange K, Dordick JS, Linhardt RJ. Heparin and anticoagulation. Front Biosci (Landmark Ed). 2016 Jun 1;21(7):1372-92. doi: 10.2741/4462. PMID 27100512
- [Result] Quaranta M, Erez O, Mastrolia SA, Koifman A, Leron E, Eshkoli T, Mazor M, Holcberg G. The physiologic and therapeutic role of heparin in implantation and placentation. PeerJ. 2015 Jan 6;3:e691. doi: 10.7717/peerj.691. eCollection 2015. PMID 25653897
- [Result] Wu XX, Guller S, Rand JH. Hydroxychloroquine reduces binding of antiphospholipid antibodies to syncytiotrophoblasts and restores annexin A5 expression. Am J Obstet Gynecol. 2011 Dec;205(6):576.e7-14. doi: 10.1016/j.ajog.2011.06.064. Epub 2011 Jun 24. PMID 21871597
- [Result] Osadchy A, Ratnapalan T, Koren G. Ocular toxicity in children exposed in utero to antimalarial drugs: review of the literature. J Rheumatol. 2011 Dec;38(12):2504-8. doi: 10.3899/jrheum.110686. Epub 2011 Oct 15. PMID 22002012